CLINICAL TRIAL: NCT06955546
Title: Probiotics And Ozonated Olive Oil To Maintain Oral Eubiosis In Stage I And II Periodontitis Patients: A Randomized, Triple-Blind Clinical Trial
Brief Title: Probiotics And Ozonated Olive Oil To Maintain Oral Eubiosis In Stage I And II Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massimo Corsalini (Other)
Responsible Party: Sponsor-Investigator, Massimo Corsalini, Associate Professor, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Organization: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Prot. 1983/CEL
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Disease; Periodontal Disease Stage 2
Keywords: periodontitis; probiotics; oral health; ozonated olive oil
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: 3 parallel arms interventional study model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Placebo Group (Placebo Comparator): In this group the patients received a placebo toothpaste, mouthwash and probiotics. Their appearance was kept identical to mimic the real products containing effective substances, in order to dissuade the patient to drop out.
  Interventions: Other: Placebo
- Group B: effective toothpaste and mouthwash. Placebo probiotics (Experimental): The patients of this group received effective toothpaste and mouthwash. Probiotics tablets were placebo.
  Interventions: Drug: Toothpaste Product; Drug: Mouthwash Product
- Group C: effective toothpaste, mouthwash and probiotics. (Experimental): The patients of this group received effective toothpaste, mouthwash and probiotics.
  Interventions: Drug: Toothpaste Product; Drug: Mouthwash Product; Dietary Supplement: Probiotic

INTERVENTIONS:
Drug: Toothpaste Product — Patients have to use the Curasept Prevent Toothpaste daily, during their domiciliar oral hygiene maneuvers.
  Link at: https://curaseptspa.it/prodotti/curasept-prevent-dentifricio/
  Other Names: Curasept Prevent Toothpaste
  Arms: Group B: effective toothpaste and mouthwash. Placebo probiotics; Group C: effective toothpaste, mouthwash and probiotics.
Drug: Mouthwash Product — Patients have to use the Curasept Prevent Mouthwash daily, during their domiciliar oral hygiene maneuvers.
  Link at: https://curaseptspa.it/prodotti/curasept-prevent-collutorio/
  Other Names: Curasept Prevent Mouthwash
  Arms: Group B: effective toothpaste and mouthwash. Placebo probiotics; Group C: effective toothpaste, mouthwash and probiotics.
Dietary Supplement: Probiotic — Patients received a daily tablet of Curasept Prevent Probiotics. Link at: https://curaseptspa.it/prodotti/curasept-prevent-probiotico-integratore-alimentare/
  Other Names: Curasept Prevent Probiotic
  Arms: Group C: effective toothpaste, mouthwash and probiotics.
Other: Placebo — Patients received a placebo toothpaste, mouthwash and probiotics. Their appearance was kept identical to mimic the real products containing effective substances, in order to dissuade the patient to drop out.
  Arms: Group A: Placebo Group

SUMMARY:
The goal of this clinical trial is to investigate the clinical benefits of the combined use of ozonized olive oil products (mouthwash and toothpaste) and probiotics on the health status of patients with Stage I and II periodontitis; could include any of the following:

* Male or female, aged between 18 and 70 years of any race.
* Diagnosis of stage I or II periodontitis according to the American Academy of Periodontology and the European Federation of Periodontology 2017 classification of periodontal diseases.
* Good general health.
* Ability to understand and comprehend the study's instructions and sign the informed consent.

The main question it aims to answer is: the single or combined use of ozonized olive oil products (mouthwash and toothpaste) and probiotics could improve the oral health status of patients with Stage I and II periodontitis compared to placebo?

Participants will proceed to their daily domiciliar oral hygiene maneuvers with the products given by investigators. The toothpaste was used twice daily, morning and evening, followed by rinsing with undiluted mouthwash for one minute. After rinsing, the patient did not rinse further with water and refrained from eating, drinking, and smoking for at least one hour. Domiciliary mechanical and drug therapies were continued, without modification, for 30 days. Moreover, the patients received a probiotic tablet daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 and 70 years of any race.
* Diagnosis of stage I or II periodontitis according to the American Academy of Periodontology and the European Federation of Periodontology 2017 classification of periodontal diseases.
* Good general health.
* Ability to understand and comprehend the study's instructions and sign the informed consent.

Exclusion Criteria:

* Pregnancy and breastfeeding.
* Periodontal or antibiotic therapy in the last two months.
* Systemic diseases that could influence the severity of periodontal disease or therapeutic success (e.g., Down syndrome, HIV, Diabetes Mellitus).
* Smoking > 10 cigarettes per day.
* Need for antibiotic prophylaxis for dental procedures.
* Chronic use of anti-inflammatory drugs, calcium channel blockers, antidepressants, and anticonvulsants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth | From enrollment to the end of treatment at 30 days
  the depth of the pocket at four sites per tooth, measured from the free gingival margin to the base of the pocket using a UNC15 periodontal probe. Periodontal pockets were classified as moderate (PPD = 4-6 mm) or deep (PPD ≥ 7 mm).
Full Mouth Plaque Score | From enrollment to the end of treatment at 30 days
  A percentage indices based on dichotomous recordings (absence/presence of plaque) recorded at four sites for each tooth present in the patient's mouth, evaluating the patient's oral hygiene status. 0% indicates the absence of plaque recorded at four sites for each tooth present in the patient's mouth, which is the best outcome possible. 100% indicates the constant presence of plaque recorded at four sites for each tooth present in the patient's mouth, which is the worst outcome possible.
Full Mouth Bleeding Score | From enrollment to the end of treatment at 30 days
  A percentage indices based on dichotomous recordings (absence/presence of bleeding) recorded at four sites for each tooth present in the patient's mouth, evaluating the patient's inflammation status. 0% indicates the absence of bleeding recorded at four sites for each tooth present in the patient's mouth, which is the best outcome possible. 100% indicates the constant presence of bleeding recorded at four sites for each tooth present in the patient's mouth, which is the worst outcome possible.

SECONDARY OUTCOMES:
Adherence | From enrollment to the end of treatment at 30 days
  The quality of adherence to the prescribed therapies was verified at each visit interval. Adherence was assessed as "valid" or "invalid."

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD about the arms and their relative outcomes could be shared, respecting the patient's privacy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From today to the next year (25/4/2026)

REFERENCES:
- See also: Curasept Prevent Mouthwash — https://curaseptspa.it/prodotti/curasept-prevent-collutorio/
- See also: Curasept Prevent Probiotics — https://curaseptspa.it/prodotti/curasept-prevent-probiotico-integratore-alimentare/
- See also: Curasept Prevent Toothpaste — https://curaseptspa.it/prodotti/curasept-prevent-dentifricio/